CLINICAL TRIAL: NCT07322003
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Pridopidine in Participants With Amyotrophic Lateral Sclerosis
Brief Title: Pridopidine Phase 3 Study to Evaluate Efficacy and Safety in ALS
Acronym: PREVAiLS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prilenia (Industry)
Collaborators: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PL101-ALS301 / FNP254-CT-2501
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — pridopidine

STUDY DESIGN:
Intervention Model Description: Randomized (3:2), double-blind, placebo-controlled study followed by an open-label extension period. During the open-label extension, all participants will receive pridopidine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pridopidine (Experimental): Pridopidine hard gelatin capsules of 45 mg strength. During titration period 1 capsule taken orally in the morning for 2 weeks. During the main treatment period, 1 capsule in the morning and 1 capsule in the afternoon taken orally. Total daily dose of 90 mg.
  Interventions: Drug: Pridopidine
- Placebo (Placebo Comparator): Placebo hard gelatin capsules. During titration period 1 capsule taken orally in the morning for 2 weeks. During the main treatment period, 1 capsule in the morning and 1 capsule in the afternoon taken orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pridopidine — Pridopidine hard gelatin capsule.
  Arms: Pridopidine
Drug: Placebo — Placebo hard gelatin capsule.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the drug pridopidine works to treat amyotrophic lateral sclerosis in adults. It will also help to learn about the safety of pridopidine. The main question it aims to answer is:

Does pridopidine slow disease progression of ALS?

Researchers will compare pridopidine to a placebo (a look-alike substance that contains no drug) to see if pridopidine works to treat ALS.

Participants will:

Take pridopidine or a placebo by mouth every day for 48 weeks. Afterwards, all participants will take pridopidine for another 48 weeks.

Visit the clinic once every 1-3 months for checkups and tests

DETAILED DESCRIPTION:
This is a Phase 3, randomized study consisting of a double-blind placebo-controlled (DBPC) period followed by an open-label extension (OLE) to evaluate the efficacy and safety of pridopidine administered orally at a dose of 45 mg twice a day in adult participants with early and rapidly progressing ALS. Standard of care treatments (e.g. riluzole, edaravone and Nuedexta) will be allowed as long as participants are on a stable dose for at least 4 weeks prior to dosing. In the DBPC period, participants will be randomized in a 3:2 ratio to the pridopidine and placebo arms.

In the DBPC period, participants will receive pridopidine or placebo for 48 weeks. In the OLE period, all participants will receive pridopidine for 48 weeks, while maintaining the blind to their original randomization for both the participant as well as the Investigator and other clinical staff. The total study duration per participant will be 102 weeks including screening and follow up.

Throughout the study, participants will be assessed through on-site clinic visits and virtual visits (via telephone).

ELIGIBILITY:
Key Inclusion Criteria:

* Definite ALS or Probable ALS using the El Escorial criteria.
* Symptom onset of ≤18 months at screening.
* Slow vital capacity (SVC) greater or equal to 60% predicted.
* Treatment Research Initiative to Cure ALS (TRICALS) Risk Profile Calculator score, based on the European Network for the Cure of ALS (ENCALS) survival prediction model, in the range of -6 to -2, inclusive, at screening.
* Able to swallow a capsule.

Key Exclusion Criteria:

* Presence of tracheostomy or permanent assisted ventilation.
* Clinically significant heart disease, clinically significant history of arrhythmia, symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia, or presence of left bundle branch block.
* Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the participant to provide informed consent and participate in the study.
* Clinically significant and/or unstable medical condition (other than ALS) that may either pose a clinically meaningful risk to the participant and/or to study completion.
* Use of medications that prolong QT interval.
* Previous treatment with pridopidine, gene therapy, or antisense oligonucleotides.
* Confirmed mutation in the SOD1, FUS or C9orf72 gene.
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline through Week 26 and Week 48 in the Revised ALS Functional Rating Scale (ALSFRS-R) total score adjusted for mortality | Baseline to Week 48
  The ALSFRS-R encompasses 12 questions grouped into 4 domains to assess bulbar symptoms, limb and trunk functionality, respiratory symptoms, and the need for percutaneous endoscopic gastrostomy (PEG), non-invasive ventilation, or tracheostomy with invasive ventilation. Each function is scored from 0 (no ability) to 4 (normal), with a minimum total score of 0 and maximum total score of 48. Higher scores indicate better functioning.

SECONDARY OUTCOMES:
Overall survival at Week 96 | Baseline to Week 96
  Time to death in days from baseline as assessed at the end of open-label extension (OLE) period
Change from baseline through Week 26 and Week 48 in speaking rate as measured by quantitative speech assessment in the clinic | Baseline to Week 48
Change from baseline through Week 48 in intelligibility of speech by quantitative speech assessment in the clinic. | Baseline to Week 48.
Change from baseline through Week 48 in percent predicted slow vital capacity (SVC) | Baseline to Week 48
  SVC measures the maximal amount of air exhaled in a relaxed expiration from full inspiration to residual volume. SVC is assessed in the sitting position with a spirometer.
Change from baseline through Week 48 in the Bulbar subdomain of the ALSFRS-R | Baseline to Week 48
  Measures decline in bulbar function.
Change from baseline through Week 48 in the Amyotrophic Lateral Sclerosis Assessment Questionnaire - 40 (ALSAQ-40) | Baseline to Week 48
  ALSAQ-40 includes 40 items/questions with 5 discrete scales including physical mobility (10 items), activities of daily living and independence (10 items), eating and drinking (3 items), communication (7 items), and emotional reactions (10 items). The questions refer to two weeks prior to the day of the application and the answers are given according to the following variables: never, rarely, sometimes, frequently and always. The score ranges from 0 to 100; the higher the score, the worse the quality of life.